CLINICAL TRIAL: NCT06853340
Title: Impact of Vascular Calcification and CASR Expression by Monocytes in Septic Shock
Acronym: CASRCHOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PI2023_843_0034
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock; Calcium Sensing Receptor; Calcium Phosphate Disorders; Inflammation; Monocyte
Keywords: Septic shock; Calcium Sensing Receptor; Calcium Phosphate disorders; Inflammation; Monocyte
MeSH Terms: conditions — Shock, Septic; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- healthy volunteers (Active Comparator)
- patients in septic shock (Experimental)
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — Patients with septic shock will have three differents times of blood sampling and of clinical and biological statements. Healthy volunteers will have a unique visit to collect clinical data and blood samples.
  Arms: patients in septic shock

SUMMARY:
In septic shock, bacterial LPS is able to activate the CaSR of cardiomyocytes inducing their apoptosis in vitro. CaSR activation in monocytes is responsible for activation of the NLRP3 inflammasome and macropinocytosis. In front of this immune axis, a variation in the monocyte expression of the CaSR is expected in the state of shock. This is already observed in other pathologies such as renal failure or in animal models of severe burns. If this is considered as an overall reflection of CaSR expression in the body, it would be consistent with the phosphocalcic disturbances associated with septic shock. The phosphocalcic balance is often modified, and not treated during the acute episode, with in particular hypocalcaemia which could be consecutive to a hyperactivation or overexpression of the CaSR. This study proposes to explore for the first time the expression of monocytic CaSR in patients in a state of shock, with possible therapeutic perspectives by the existence of calcimimetics and calcilytics. In this study, the investigators propose to explore the CasR and its implication in septic shock in a three - part protocol : measurement by flow cytometry of monocyte expression of CASR (primary objective) and CD33, CD14, CD163, CD16 and HLA-DR), survey of clinical and biological parameters in patients with septic shock and healthy volunteers and acquisition of calcium score in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over the age of 18,
* patients who have not participated in a study evaluating an investigational drug in the 30 days preceding the samples,
* intensive care patients in a state of septic shock within the first 24 hours of the introduction of pressor amines,
* French resident year-round,
* lactate > 2mmol/L,
* patients with social security coverage.

Exclusion Criteria:

* Patients in hemorrhagic shock,
* history of parathyroidectomy, patient with hypersecretion of PTHrp,
* sarcoidosis,
* genetic disturbance of CaSR including familial hypocalciuric hypercalcaemia,
* current immunosuppressant treatment (anticalcineurin, mTOR inhibitor, methotrexate, high-dose corticosteroids excluding hydrocortisone and fludrocortisone),
* chronic myelomonocytic leukemia,
* patients with febrile neutropenia,
* patients with acquired or constitutional immune system,
* pregnant or breastfeeding patient,
* patients under curators, guardianship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Monocyte CaSR expression in healthy patient | 1 day
  Monocyte CaSR expression in healthy patient

SECONDARY OUTCOMES:
Monocyte CasR expression in patient with septic shock | day 0
  Monocyte CasR expression in patient with septic shock
Monocyte CasR expression in patient with septic shock | day 2
  Monocyte CasR expression in patient with septic shock
Monocyte CasR expression in patient with septic shock | day 7
  Monocyte CasR expression in patient with septic shock

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No